CLINICAL TRIAL: NCT02209610
Title: Premature Fatigue in Veterans With Heart Failure: Neuronal Influences
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: E1572-P
Record Dates: First submitted 2014-07-10; First posted 2014-08-06 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients With Heart Failure: Neuromuscular Abnormalities (Other): Patients with Heart Failure
  Interventions: Device: Electrical and Magnetic Nerve Stimulators; Drug: Intrathecal Fentanyl
- Health Control Subjects and Neuromuscular Function (Other): Health Control Subjects
  Interventions: Device: Electrical and Magnetic Nerve Stimulators; Drug: Intrathecal Fentanyl

INTERVENTIONS:
Device: Electrical and Magnetic Nerve Stimulators — Stimulation of motor nerve and central nervous system
Drug: Intrathecal Fentanyl — Mu-opioid receptor agonist

SUMMARY:
A hallmark of patients with heart failure (HF) is premature fatigue which impairs their quality of life and depicts a major source of morbidity. Premature fatigue may be attributed to a) contraction-induced transient changes within muscles (i.e. peripheral fatigue) and/or b) failure of the central nervous system to 'drive' / activate locomotor muscles (i.e. central fatigue). Both determinants of fatigue can lead to a reduction in a muscle's force and power generating capacity and to a compromised ability to perform whole body activities (e.g. walking). Recent findings in health have documented that group III/IV afferent fibers from the working muscle play a critical role in the development of both components of fatigue. Specifically, group III/IV muscle afferents limit central motor drive (CMD) during exercise and thereby exaggerate the development of central fatigue. In contrast, muscle afferents optimize muscle O2 delivery through the precise regulation of circulation and ventilation during exercise and thereby attenuate the development of peripheral fatigue.

DETAILED DESCRIPTION:
Recent findings in HF suggest an altered effect of group III/IV muscle afferents in this population. Although normal afferent feedback is crucial for adequate O2 delivery during exercise, excessive neural feedback has substantial negative consequences. HF patients are characterized by augmented neural feedback arising from overactive muscle afferents. It has been hypothesized that this abnormality compromises locomotor muscle O2 delivery in these patients. Therefore, the abnormally elevated muscle afferent feedback in HF might exacerbate, compared to healthy age- and activity matched individuals (CTRLs), the development of both peripheral (via limiting O2 delivery) and central (via restricting CMD) fatigue during exercise. Recent advances in non-invasive stimulation techniques offer a genuine opportunity to identify the sites and synaptic mechanisms that mediate central and peripheral fatigue including alterations in the responsiveness of the corticospinal tract (i.e. a determinant of central fatigue). Taken together, the proposed studies aim to determine the impact of HF on the precise development of central and peripheral fatigue during both whole body and single muscle exercise and evaluate the extent to which group III/IV muscle afferents contribute to this development.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a history of stable cardiomyopathy (ischemic and non-ischemic, >1yr duration, ages 20-75 yr),
* not pacemaker dependent (no biventricular pacers),
* NYHA class II and III symptoms,
* Left ventricular ejection fraction (LVEF)<35%,
* no or minimal smoking history (<15 pk yrs) and on stable medications.
* The investigators will also study subjects with preserved ejection fraction

  * heart failure with a preserved ejection fraction (HFpEF);
  * LVEF >50%,
  * >1yr duration,
  * ages 20-75 yr,
* not pacemaker dependent,
* NYHA class II and III symptoms,
* no or minimal smoking history (<15 pk yrs) and on stable medications. The investigators will exclude morbidly obese patients (BMI >35), patients with uncontrolled hypertension (>160/100), anemia (Hgb<9) and severe renal insufficiency (individuals with creatinine clearance <30 by the Cockcroft-Gault formula).

Exclusion Criteria:

* Patients with significant non-cardiac comorbidities, which if present could alter the study results, will be excluded.
* Patients will be sedentary, defined here as no regular physical activity for at least the prior 6 months and current activity level will be documented by an activity questionnaire.
* Candidates must have no orthopedic limitations that would prohibit them from performing exercise.
* Due to the typical age of patients with heart failure, all women will be postmenopausal (either natural or surgical) defined as a cessation of menses for at least 2 years,

  * and in women without a uterus, follicle stimulating hormone (FSH) >40 IU/L.
* Women currently taking hormone replacement therapy (HRT) will be excluded from the proposed studies due to the direct vascular effects of HRT.
* Patients with a pacemaker and / or defibrillator will be excluded from the study due to the use of a magnetic/electric stimulators.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Amann, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ives SJ, Amann M, Venturelli M, Witman MA, Groot HJ, Wray DW, Morgan DE, Stehlik J, Richardson RS. The Mechanoreflex and Hemodynamic Response to Passive Leg Movement in Heart Failure. Med Sci Sports Exerc. 2016 Mar;48(3):368-76. doi: 10.1249/MSS.0000000000000782. PMID 26418560
- [Result] Sidhu SK, Weavil JC, Venturelli M, Rossman MJ, Gmelch BS, Bledsoe AD, Richardson RS, Amann M. Aging alters muscle reflex control of autonomic cardiovascular responses to rhythmic contractions in humans. Am J Physiol Heart Circ Physiol. 2015 Nov;309(9):H1479-89. doi: 10.1152/ajpheart.00433.2015. Epub 2015 Sep 18. PMID 26386110
- [Result] Weavil JC, Sidhu SK, Mangum TS, Richardson RS, Amann M. Fatigue diminishes motoneuronal excitability during cycling exercise. J Neurophysiol. 2016 Oct 1;116(4):1743-1751. doi: 10.1152/jn.00300.2016. Epub 2016 Jul 20. PMID 27440242
- [Result] Amann M, Sidhu SK, Weavil JC, Mangum TS, Venturelli M. Autonomic responses to exercise: group III/IV muscle afferents and fatigue. Auton Neurosci. 2015 Mar;188:19-23. doi: 10.1016/j.autneu.2014.10.018. Epub 2014 Oct 23. PMID 25458423
- [Result] Wray DW, Amann M, Richardson RS. Peripheral vascular function, oxygen delivery and utilization: the impact of oxidative stress in aging and heart failure with reduced ejection fraction. Heart Fail Rev. 2017 Mar;22(2):149-166. doi: 10.1007/s10741-016-9573-4. PMID 27392715

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Heart Failure: Neuromuscular Abnormalities: Patients with Heart Failure are characterized by excessive exercise-induced neuromuscular fatigue Electrical and Magnetic Nerve Stimulators: Stimulation of motor nerve and central nervous system
  Intrathecal Fentanyl: Mu-opioid receptor agonist
Period: Overall Study
Arm/Group | Patients With Heart Failure: Neuromuscular Abnormalities | Health Control Subjects and Neuromuscular Function
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Heart Failure: Neuromuscular Abnormalities | Health Control Subjects and Neuromuscular Function | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (3) | 64 (3) | 66 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximal Voluntary Quadriceps Force [% Change From Baseline]
Description: Following dynamic single leg knee extension exercise for a given duration (4-8 min), the decline in maximal voluntary contraction force will be measured.
Time Frame: 1 minute after exercise on study day
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Patients With Heart Failure: Neuromuscular Abnormalities | Health Control Subjects and Neuromuscular Function
Number analyzed (Participants) | 16 | 16
percentage change | -30 (3) | -5 (2)

2. Primary Outcome: Quadriceps Twitch Force and Voluntary Activation (% Change From Baseline)
Description: During a 2-min maximal voluntary quadriceps contraction, central and peripheral fatigue will develop progressively and significantly more in HF vs. CTRLs.
Time Frame: During (20 second intervals) and 1 minute after exercise on study day
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Patients With Heart Failure: Neuromuscular Abnormalities | Health Control Subjects and Neuromuscular Function
Number analyzed (Participants) | 16 | 16
percentage change
  Twitch force | -60 (5) | -35 (6)
  Voluntary activation [VA] | -25 (6) | -20 (5)

3. Primary Outcome: Muscle Afferent Affect
Description: Corticospinal responsiveness will be quantified before and after exercise.
Time Frame: 1 minute after exercise on study day
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Patients With Heart Failure: Neuromuscular Abnormalities | Health Control Subjects and Neuromuscular Function
Number analyzed (Participants) | 16 | 16
percent change | -30 (3) | 10 (8)

ADVERSE EVENTS:
Arm/Group | Patients With Heart Failure: Neuromuscular Abnormalities | Health Control Subjects and Neuromuscular Function
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No